CLINICAL TRIAL: NCT00507507
Title: A Randomized, Double-Blind Study Evaluating Tenofovir Disoproxil Fumarate (DF) Monotherapy Versus the Combination of Emtricitabine and Tenofovir DF for the Treatment of Chronic Hepatitis B
Brief Title: A Study to Compare Tenofovir DF Versus the Combination of Emtricitabine Plus Tenofovir DF for the Treatment of Chronic Hepatitis B in Patients With Normal Alanine Aminotransferase (ALT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-203-0101
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Hepatitis B
Keywords: tenofovir; monotherapy; emtricitabine; combination; hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir DF (Experimental): Participants were randomized to receive tenofovir DF plus placebo to match FTC once daily.
  Interventions: Drug: Tenofovir DF; Drug: Placebo
- FTC+Tenofovir DF (Experimental): Participants were randomized to receive FTC plus tenofovir DF once daily.
  Interventions: Drug: Tenofovir DF; Drug: FTC

INTERVENTIONS:
Drug: Tenofovir DF — Tenofovir disoproxil fumarate (tenofovir DF) 300 mg tablet taken orally once daily
  Other Names: Viread®
Drug: FTC — Emtricitabine (FTC) 200 mg capsule taken orally once daily
  Other Names: Emtriva®
  Arms: FTC+Tenofovir DF
Drug: Placebo — Placebo to match FTC taken once daily
  Arms: Tenofovir DF

SUMMARY:
The main objective of the study was to evaluate the antiviral activity of tenofovir disoproxil fumarate (tenofovir DF) monotherapy versus emtricitabine (FTC) plus tenofovir DF combination therapy for the treatment of chronic hepatitis B (HBV) in participants in the immune tolerant phase of HBV infection.

The efficacy of tenofovir DF monotherapy versus FTC plus tenofovir DF combination therapy was evaluated for suppression of the virus (decrease in HBV DNA), serological response (generation of antibodies to the virus), biochemical response (changes in liver enzymes), and the development of drug-resistant mutations. The safety and tolerability of both tenofovir DF monotherapy and FTC plus tenofovir DF were evaluated by routine monitoring for adverse events and changes in laboratory parameters.

Participants were randomized in a 1:1 ratio to receive tenofovir DF monotherapy or FTC plus tenofovir DF. All subjects were to continue on blinded study medication until the last subject reached Week 192. Participants who permanently discontinued study drug (on or before Week 192) were followed for a 24-week treatment-free follow-up period, or until initiation of alternative HBV therapy, whichever occurred first. Subjects who discontinued study drug on or after Week 48 because of hepatitis B surface antigen (HBsAg) loss or seroconversion to antibody to hepatitis B surface antigen (anti-HBs), however, were to have returned for their regularly scheduled through Week 192 and every 16 weeks thereafter until the last subject reached Week 192.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection, defined as positive serum HBsAg for at least 6 months or HBsAg positive > 3 months and positive for immunoglobulin G antibody against hepatitis B core antigen
* 18 through 69 years of age, inclusive
* Hepatitis B e antigen (HBeAg) positive
* HBV DNA ≥ 10^8 copies/mL
* ALT ≤ the upper limit of the normal range (ULN)
* Willing and able to provide written informed consent
* Negative serum beta-human chorionic gonadotropin (for females of childbearing potential only)
* Calculated creatinine clearance ≥ 70 mL/min
* Hemoglobin ≥ 10 g/dL
* Neutrophils ≥ 1,500/mm^3
* No prior oral HBV therapy (eg, nucleotide and/or nucleoside therapy or other investigational agents for HBV infection)

Exclusion Criteria:

* Pregnant women, women who were breast feeding, or who believed they may have wished to become pregnant during the course of the study
* Males and females of reproductive potential unwilling to use an effective method of contraception during the study
* Decompensated liver disease defined as direct (conjugated) bilirubin > 1.2 x ULN, prothrombin time > 1.2 x ULN, platelets < 150,000/mm^3, serum albumin < 3.5 g/dL, or prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, or variceal hemorrhage)
* Received interferon (pegylated or not) therapy within 6 months of the screening visit
* Alpha-fetoprotein > 50 ng/mL
* Evidence of hepatocellular carcinoma
* Coinfection with hepatitis C virus (by serology), HIV, or hepatitis D virus
* Significant renal, cardiovascular, pulmonary, or neurological disease
* Received solid organ or bone marrow transplantation
* Was currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion
* Had proximal tubulopathy
* Known hypersensitivity to the study drugs, the metabolites, or formulation excipients

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-09; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (9):
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Miami, Florida
  - Detroit, Michigan
  - Manhasset, New York
  - New York, New York
  - Germantown, Tennessee
  - Seattle, Washington
- Australia (4):
  - Camperdown, New South Wales
  - Westmead, New South Wales
  - Heidelburg, Victoria
  - Melbourne, Victoria
- Canada (3):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
- France (3):
  - Lille
  - Lyon
  - Strasbourg
- Germany (8):
  - Berlin
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Mainz
- Hong Kong (3):
  - Pokfulam
  - Shatin
  - Tai Po
- New Zealand (2):
  - Grafton, Auckland
  - Hamilton
- Poland (3):
  - Bydgoszcz
  - Chorzów
  - Warsaw
- Singapore, Singapore
- Taiwan (4):
  - Kaohsiung City
  - Kaoshiung
  - Tainan
  - Taipei
- United Kingdom (2):
  - London
  - Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 34 sites in the North America, Europe, Asia, Australia, and New Zealand. The first participant was screened on 04 September 2007. The last participant observation for the Week 192 analysis was on 03 February 2012.
Pre-assignment Details: 309 participants were screened and 129 were randomized; 126 randomized participants received at least one dose of study drug, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- Tenofovir DF: Participants were randomized to receive tenofovir disoproxil fumarate (tenofovir DF; 300 mg tablet) plus placebo to match emtricitabine (FTC; tablet) orally once daily.
- FTC+Tenofovir DF: Participants were randomized to receive FTC (200 mg tablet) plus tenofovir DF (300 mg tablet) orally once daily.
Period: Treatment Period
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Started | 64 | 62
Completed 192 Weeks of Treatment | 52 | 52
Completed | 12 | 9
Not Completed | 52 | 53
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 4 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 46 | 47
Period: 24-week Treatment-free Follow-up Period
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Started | 26 (Participants who discontinued treatment early may have entered the treatment-free follow-up period.) | 29 (Participants who discontinued treatment early may have entered the treatment-free follow-up period.)
Completed | 16 | 12
Not Completed | 10 | 17
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 9 | 16

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and treated were analyzed for baseline characteristics.
Groups:
- Tenofovir DF: Participants were randomized to receive tenofovir DF (300 mg tablet) plus placebo to match FTC (tablet) orally once daily.
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | FTC+Tenofovir DF | Total
Number analyzed (Participants) | 64 | 62 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9.5) | 33 (11.2) | 33 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 31 | 31 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 64 | 62 | 126
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 56 | 56 | 112
  White | 4 | 1 | 5
  Black | 2 | 2 | 4
  Pacific Islander | 1 | 3 | 4
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment. (Tenofovir DF, n = 65; FTC+tenofovir DF, n = 64.)
  participants
    Australia | 0 | 2 | 2
    Canada | 4 | 3 | 7
    France | 4 | 3 | 7
    Germany | 3 | 3 | 6
    Hong Kong | 28 | 33 | 61
    New Zealand | 2 | 4 | 6
    Poland | 2 | 0 | 2
    Singapore | 2 | 0 | 2
    Taiwan | 6 | 6 | 12
    United Kingdom | 0 | 2 | 2
    United States | 14 | 8 | 22
Hepatitis B Virus (HBV) DNA [Mean (Standard Deviation); unit: log_10 copies/mL] | 9.18 (0.402) | 9.16 (0.395) | 9.17 (0.397)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 26.9 (14.05) | 26.2 (9.88) | 26.6 (12.13)
Hepatitis B e Antigen (HBeAg) [Number; unit: participants]
  Negative | 1 | 0 | 1
  Positive | 63 | 62 | 125
Antibody to HBeAg (Anti-HBe) [Number; unit: participants]
  Negative | 0 | 1 | 1
  Positive | 1 | 0 | 1
  Missing/Unevaluable | 63 | 61 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Week 192
Description: The percentage of participants with HBV DNA < 400 copies/mL at Week 192 was analyzed. Participants with missing data were considered to have failed to achieve the criteria for evaluation.
Time Frame: Week 192
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
percentage of participants | 54.7 | 75.8
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; The null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 400 copies/mL at Week 192 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference. The sample size provided at least 85% power to detect a difference of 30% between the groups, assuming response rates of 30% and 60% in the Tenofovir DF and FTC+Tenofovir DF groups, respectively; Test type: Superiority or Other; p = 0.016, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used

2. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Weeks 48, 96, and 144
Description: The percentage of participants with HBV DNA < 400 copies/mL at Weeks 48, 96, and 144 was analyzed. Participants with missing data were considered to have failed to achieve the criteria for evaluation.
Time Frame: Weeks 48, 96, and 144
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
percentage of participants
  Week 48 | 40.6 | 59.7
  Week 96 | 53.1 | 75.8
  Week 144 | 62.5 | 80.6
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 48: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 400 copies/mL at Week 48 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.050, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 2: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 96: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 400 copies/mL at Week 96 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.009, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 3: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 144: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 400 copies/mL at Week 144 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.030, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used

3. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL at Weeks 48, 96, 144, and 192
Description: The percentage of participants with HBV DNA < 169 copies/mL at Weeks 48, 96, 144, and 192 was analyzed. Participants with missing data were considered to have failed to achieve the criteria for evaluation.
Time Frame: Weeks 48, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
percentage of participants
  Week 48 | 29.7 | 33.9
  Week 96 | 45.3 | 64.5
  Week 144 | 50.0 | 72.6
  Week 192 | 45.3 | 69.4
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 48: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 169 copies/mL at Week 48 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.703, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 2: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 96: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 169 copies/mL at Week 96 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.034, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 3: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 144: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 169 copies/mL at Week 144 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.011, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 4: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 192: the null hypothesis was that there was no difference in the proportion of subjects with HBV DNA < 169 copies/mL at Week 192 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.007, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used

4. Secondary Outcome: Change From Baseline in HBV DNA at Week 48
Description: The change from baseline in HBV DNA at Week 48 was analyzed.
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with evaluable change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 58
log_10 copies/mL | -6.22 (0.608) | -6.49 (0.577)
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; The null hypothesis was that there was no difference of change in HBV DNA from baseline between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — A Wilcoxon rank-sum (2-sided) test was used, with no adjustments for covariates

5. Secondary Outcome: Change From Baseline in HBV DNA at Week 96
Description: The change from baseline in HBV DNA at Week 96 was analyzed.
Time Frame: Baseline to Week 96
Population: Participants in the Full Analysis Set with evaluable change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 59 | 56
log_10 copies/mL | -6.46 (0.763) | -6.55 (1.176)
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney) — A Wilcoxon rank-sum (2-sided) test was used, with no adjustments for covariates

6. Secondary Outcome: Change From Baseline in HBV DNA at Week 144
Description: The change from baseline in HBV DNA at Week 144 was analyzed.
Time Frame: Baseline to Week 144
Population: Participants in the Full Analysis Set with evaluable change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 55 | 56
log_10 copies/mL | -6.66 (0.655) | -6.62 (1.318)
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.186, Wilcoxon (Mann-Whitney) — A Wilcoxon rank-sum (2-sided) test was used, with no adjustments for covariates

7. Secondary Outcome: Change From Baseline in HBV DNA at Week 192
Description: The change from baseline in HBV DNA at Week 192 was analyzed.
Time Frame: Baseline to Week 192
Population: Participants in the Full Analysis Set with evaluable change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 53 | 54
log_10 copies/mL | -6.32 (1.463) | -6.70 (0.913)
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.070, Wilcoxon (Mann-Whitney) — A Wilcoxon rank-sum (2-sided) test was used, with no adjustments for covariates

8. Secondary Outcome: Number of Participants With Normal Alanine Aminotransferase (ALT) at Weeks 48, 96, 144, and 192
Description: Range of normal ALT was 6 to 34 U/L for females, 6 to 43 U/L for males. Participants with missing data were considered to have failed to achieve the criteria for evaluation.
Time Frame: Weeks 48, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
participants
  Week 48 | 52 | 54
  Week 96 | 52 | 50
  Week 144 | 51 | 46
  Week 192 | 41 | 44
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 48: the null hypothesis was that there was no difference in the proportion of subjects with normal ALT at Week 48 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.467, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used, with no adjustments for covariates
Statistical Analysis 2: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 96: the null hypothesis was that there was no difference in the proportion of subjects with normal ALT at Week 96 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 1.000, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used, with no adjustments for covariates
Statistical Analysis 3: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 144: the null hypothesis was that there was no difference in the proportion of subjects with normal ALT at Week 144 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.529, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used, with no adjustments for covariates
Statistical Analysis 4: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 192: the null hypothesis was that there was no difference in the proportion of subjects with normal ALT at Week 192 between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.451, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used, with no adjustments for covariates

9. Secondary Outcome: Number of Participants With Hepatitis B e Antigen (HBeAg) Loss at Weeks 48, 96, 144, and 192
Description: The number of participants with HBeAg loss at Weeks 48, 96, 144, and 192 was analyzed. Loss of HBeAg was defined as change of detectable HBeAg from positive to negative.
  No statistical analysis is presented for Week 48 because no participants met the criteria at that time point.
Time Frame: Weeks 48, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg positive at baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 63 | 62
participants
  Week 48 | 0 | 0
  Week 96 | 2 | 0
  Week 144 | 4 | 0
  Week 192 | 4 | 1
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 96: the null hypothesis was that there was no difference in the proportion of subjects with HBeAg loss between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.496, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 2: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 144: the null hypothesis was that there was no difference in the proportion of subjects with HBeAg loss between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.119, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 3: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 192: the null hypothesis was that there was no difference in the proportion of subjects with HBeAg loss between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.365, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used

10. Secondary Outcome: Number of Participants With Seroconversion to Antibody Against HBeAg (Anti-HBe) at Weeks 48, 96, 144, and 192
Description: The number of participants with seroconversion to anti-HBe at Weeks 48, 96, 144, and 192 was analyzed. Seroconversion to anti-HBe was defined as change of detectable antibody to HBeAg from negative to positive.
  No statistical analysis is presented for Week 48 because no participants met the criteria at that time point.
Time Frame: Weeks 48, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg positive at baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 63 | 62
participants
  Week 48 | 0 | 0
  Week 96 | 2 | 0
  Week 144 | 4 | 0
  Week 192 | 3 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 96: the null hypothesis was that there was no difference in the proportion of subjects with seroconversion to anti-HBe between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.496, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 2: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 144: the null hypothesis was that there was no difference in the proportion of subjects with seroconversion to anti-HBe between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.119, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used
Statistical Analysis 3: Comparison: Tenofovir DF vs FTC+Tenofovir DF; Analysis at Week 192: the null hypothesis was that there was no difference in the proportion of subjects with seroconversion to anti-HBe between the Tenofovir DF and FTC+Tenofovir DF groups; the alternative hypothesis was that there was a difference; Test type: Superiority or Other; p = 0.244, Fisher Exact — A Fisher exact test with a 0.05 two-sided significance level was used

11. Secondary Outcome: Number of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Weeks 48, 96, 144, and 192
Description: The number of participants with HBsAg loss at Weeks 48, 96, 144, and 192 was analyzed. Loss of HBsAg was defined as change of detectable HBsAg from positive to negative.
Time Frame: Weeks 48, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
participants
  Week 48 | 0 | 0
  Week 96 | 0 | 0
  Week 144 | 0 | 0
  Week 192 | 0 | 0

12. Secondary Outcome: Number of Participants With Seroconversion to Antibody to HBsAg (Anti-HBs) at Weeks 48, 96, 144, and 192
Description: The number of participants with seroconversion to anti-HBs at Weeks 48, 96, 144, and 192 was analyzed. Seroconversion to anti-HBs was defined as change of detectable antibody to HBsAg from negative to positive.
Time Frame: Weeks 48, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 64 | 62
participants
  Week 48 | 0 | 0
  Week 96 | 0 | 0
  Week 144 | 0 | 0
  Week 192 | 0 | 0

13. Secondary Outcome: Occurrence of HBV Resistance Mutations
Description: The development of HBV resistance mutations (occurrence of conserved site changes and/or polymorphic site changes) was analyzed for the overall study period (through Week 192).
Time Frame: Baseline to Week 192
Population: Genotyping was attempted for all participants with HBV DNA ≥ 400 copies/mL at Week 48, 96, 144, 192 and/or the early discontinuation visit, and for all participants (with HBV DNA ≥ 400 copies/mL) after Week 192 who were on study for at least 216 weeks when the last participant reached Week 192.
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC+Tenofovir DF
Number analyzed (Participants) | 40 | 29
participants
  Conserved (with/without polymorphic) site changes | 6 | 5
  Polymorphic site changes only | 16 | 9

ADVERSE EVENTS:
Time Frame: Baseline until the last participant reached Week 192, and 24-week treatment-free follow-up.
Description: Treatment-emergent adverse events were collected until the last participant reached Week 192.
  Adverse events were also collected for those participants who permanently discontinued study drug on or before Week 192 and were followed for 24 weeks off treatment or until initiation of alternative HBV therapy, whichever occurred first.
Groups:
- Tenofovir DF (Treatment Period): Participants were randomized to receive tenofovir DF (300 mg tablet) plus placebo to match FTC (tablet) orally once daily.
  Adverse events (AEs) for this reporting group are reported for the entire treatment period.
- FTC+Tenofovir DF (Treatment Period): Participants were randomized to receive FTC (200 mg tablet) plus tenofovir DF (300 mg tablet) orally once daily.
  AEs for this reporting group are reported for the entire treatment period.
- Tenofovir DF (24-week Treatment-free Follow-up Period): This reporting group includes participants randomized to the Tenofovir DF group who permanently discontinued study drug on or before the last subject reached Week 192 and were followed for 24 weeks off treatment or until initiation of alternative HBV therapy, whichever occurred first.
  AEs reported for this reporting group are those that occurred during the 24-week treatment-free follow-up period only.
- FTC+Tenofovir DF (24-week Treatment-free Follow-up Period): This reporting group includes participants randomized to the FTC+Tenofovir DF group who permanently discontinued study drug on or before the last subject reached Week 192 and were followed for 24 weeks off treatment or until initiation of alternative HBV therapy, whichever occurred first.
  AEs reported for this reporting group are those that occurred during the 24-week treatment-free follow-up period only.
Arm/Group | Tenofovir DF (Treatment Period) | FTC+Tenofovir DF (Treatment Period) | Tenofovir DF (24-week Treatment-free Follow-up Period) | FTC+Tenofovir DF (24-week Treatment-free Follow-up Period)
Serious Adverse Events (participants affected / at risk) | 6/64 | 3/62 | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 41/64 | 39/62 | 2/26 | 7/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (Treatment Period) (N=64) | FTC+Tenofovir DF (Treatment Period) (N=62) | Tenofovir DF (24-week Treatment-free Follow-up Period) (N=26) | FTC+Tenofovir DF (24-week Treatment-free Follow-up Period) (N=29)
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (Treatment Period) (N=64) | FTC+Tenofovir DF (Treatment Period) (N=62) | Tenofovir DF (24-week Treatment-free Follow-up Period) (N=26) | FTC+Tenofovir DF (24-week Treatment-free Follow-up Period) (N=29)
Influenza (Infections and infestations) | 14 | 12 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 8 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 6 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Influenza like illness (General disorders) | 6 | 6 | 0 | 0
Fatigue (General disorders) | 5 | 4 | 0 | 2
Asthenia (General disorders) | 4 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 10 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years